CLINICAL TRIAL: NCT03993132
Title: Cardiovascular Outcomes, and Mortality in Danish Patients With Type 2 Diabetes Who Initiate Empagliflozin Versus Glucagon-Like Peptide-1 Receptor Agonists (GLP1-RA): A Danish Nationwide Comparative Effectiveness Study [EMPLACEtm]
Brief Title: A Study Using Medical Records of Danish People With Type 2 Diabetes Comparing Empagliflozin and Glucagon-Like Peptide-1 Receptor Agonists (GLP1-RA) in the Occurrence of Serious Cardiovascular Outcomes
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1245-0194
Record Dates: First submitted 2019-06-19; First posted 2019-06-20 (Actual); Results first posted 2024-02-12 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2023-06

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — empagliflozin; Liraglutide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other

GROUPS / COHORTS (1):
- Patients with type 2 diabetes
  Interventions: Drug: Empagliflozin; Drug: Liraglutide

INTERVENTIONS:
Drug: Empagliflozin — new users (initiators) of Empagliflozin
Drug: Liraglutide — initiators of Liraglutide

SUMMARY:
The primary research question is to evaluate whether, among patients with type 2 diabetes mellitus (T2D), initiation of empagliflozin changes the adjusted incidence of outcomes compared with initiation of Glucagon-Like Peptide-1 Receptor Agonists (GLP1-RA).

ELIGIBILITY:
Inclusion Criteria:

The empagliflozin-exposed population must also meet the following criteria:

* Have at least one prescription for empagliflozin or fixed-dose combination of empagliflozin with another drug, with or without treatment with another glucose-lowering drug
* Have no prescription/dispensing of SGLT2 inhibitors (including empagliflozin) alone or in fixed-dose combination prior to the index date
* Have no prescription/dispensing of a GLP-1 receptor agonist alone or in fixed dose combination prior to the index date

The population exposed to GLP1-RA must meet the following criteria:

* Have at least one prescription for GLP1-RA or a fixed-dose combination of GLP1-RA with another drug, with or without treatment with another glucose-lowering drug.
* Have no prescription/dispensing of a GLP-1 receptor agonist alone or in fixed dose combination prior to the index date
* Have no prescription/dispensing of SGLT2 inhibitors (including empagliflozin) alone or in fixed-dose combination prior to the index date

Exclusion Criteria:

-Patients with type 1 diabetes T1D before the index date will not be included in the study.

Exclusion criteria by outcome of interest: Different exclusion criteria will be applied to generate sets of cohorts for the analysis of the different outcomes of interest.

In one main analysis, we will assess co-primary and secondary outcomes among all patients, regardless of a history of previous outcome events being present or not. In other words, we will allow a previous history of CVD events. We will adjust for the history of these events in the regression model rather than excluding patients with previous events (e.g. assess outcome rates of myocardial infarction in empagliflozine and liraglutide initiators while adjusting for previous history of myocardial infarction, unstable angina, or coronary revascularization).

In another main analysis of outcomes, we will exclude patients who had a specific outcome previously.

For example in the analysis of the primary heart failure outcome (heart failure admission or loop-diuretics), patients will not be included if a diagnosis of heart failure is recorded any time before or at the index date, or if a prescription for loop-diuretics has been filled within 12 months before or at the index date. For the secondary outcome of acute hospital admission with heart failure, we will include also patients with previous prescription for loop-diuretics, but exclude those with previous heart failure admission.

For analysis of stroke, patients will not be included if a diagnosis of stroke is recorded any time before or at the index date.

For analysis of myocardial infarction, unstable angina, or coronary revascularization, patients will not be included if any of these 3 major atherosclerotic cardiovascular events are recorded any time before or at the index date.

In additional analyses, other criteria will apply (To be discussed, RWT). Thus, an additional analysis will include also patients with previous outcome events, and adjust for the history of these events in the regression model rather than excluding them (e.g. assess outcome rates of myocardial infarction in empagliflozine and liraglutide initiators while adjusting for previous history of myocardial infarction, unstable angina, or coronary revascularization).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The source population for our study consists of individuals with type 2 diabetes, who are defined in our study as individuals who live in Denmark and who have never used oral antihyperglycemic drugs or insulin.
Sampling Method: Non-Probability Sample
Enrollment: 26774 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2022-06-16 (Actual); Study Completion 2022-06-16 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Clinical Epidemiology - Aarhus Unversiteteshospital, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- [Derived] Thomsen RW, Christensen LWB, Kahlert J, Knudsen JS, Ustyugova A, Sandgaard S, Holmgaard P, Ehlers LH, Sorensen HT. Healthcare Resource Utilization and Costs for Empagliflozin Versus Glucagon-Like Peptide-1 Receptor Agonists in Routine Clinical Care in Denmark. Diabetes Ther. 2022 Dec;13(11-12):1891-1906. doi: 10.1007/s13300-022-01323-y. Epub 2022 Oct 31. PMID 36315384
- See also: Related Info — https://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This non-interventional cohort study based on existing data planned to compare new users of empagliflozin with new users of Glucagon-Like Peptide-1 Receptor Agonists (GLP-1RA) in Denmark between 21015 and 2020. Due to a huge shift after 2018 in drug type use within the GLP-1RA group the final analysis was not completed.
Pre-assignment Details: All subjects were screened for eligibility to ensure that they (the subjects) strictly met all inclusion and none of the exclusion criteria.
Groups:
- Empagliflozin - PS Balanced Cohort: All eligible adult patients (>18 years) with type 2 diabetes (T2D) initiating treatment with empagliflozin in Denmark between 2015 and 2018, who were included in danish population-based linked registries (Civil Registration System, Danish National Patient Register, National Database of Reimbursed Prescriptions, LABKA Database). Patients were followed-up through 2020. Propensity score (PS) balancing was applied to match new users of empagliflozin to new users of liraglutide.
- Liraglutide - PS Balanced Cohort: All eligible adult patients (>18 years) with type 2 diabetes (T2D) initiating treatment with liraglutide in Denmark between 2015 to 2018, who were included in danish population-based linked registries (Civil Registration System, Danish National Patient Register, National Database of Reimbursed Prescriptions, LABKA Database). Patients were followed-up through 2020. Propensity score (PS) balancing was applied to match new users of empagliflozin to new users of liraglutide.
Period: Overall Study
Arm/Group | Empagliflozin - PS Balanced Cohort | Liraglutide - PS Balanced Cohort
Started (Propensity score balanced cohort) | 14148 | 12626
Completed | 14148 | 12626
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All patients included in the propensity score (PS) balanced cohort of either empagliflozin or liraglutide users.
Groups:
- Total: Total of all reporting groups
Arm/Group | Empagliflozin - PS Balanced Cohort | Liraglutide - PS Balanced Cohort | Total
Number analyzed (Participants) | 14148 | 12626 | 26774
Age, Continuous [Median (Inter-Quartile Range); unit: Years] | 61.55 [52.73 to 69.83] | 61.19 [52.31 to 69.83] | 61.37 [52.54 to 69.70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5692 | 5162 | 10854
  Male | 8456 | 7464 | 15920
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Incidence Rate of Expanded Major Adverse Cardiovascular Event (MACE) Composite Outcome - OT Analysis
Description: Composite outcome includes: All-cause death, acute admission with non-fatal (within 30 days) stroke, with non-fatal (within 30 days) myocardial infarction (MI), admission with unstable angina, coronary revascularization, or acute admission with non-fatal heart failure (HF).
  The results from on-treatment (OT) analysis are reported. For the OT analyses, treatment duration was based on the estimated number of days covered by each filled prescription, calculated as the number of drug packages times the numerical volume of a package. A grace period of 30 days were added.
  In the OT analysis, participants were censored from further follow-up at either treatment cessation, initiation of an alternative drug in the study drug class and initiation of a drug from the comparator study drug class.
Time Frame: From first initiation of empagliflozin or liraglutide until end of follow-up, up to 6 years.
Population: All patients included in the propensity score (PS) balanced cohort of either empagliflozin or liraglutide users.
Measure: Number; unit: Events per 1000 person-years
Arm/Group | Empagliflozin - PS Balanced Cohort | Liraglutide - PS Balanced Cohort
Number analyzed (Participants) | 14148 | 12626
Events per 1000 person-years | 36.1 | 35.9
Statistical Analysis 1: Comparison: Empagliflozin - PS Balanced Cohort vs Liraglutide - PS Balanced Cohort; Test type: Other — A Cox regression with selected variables based on previous literature, covariate data availability, examination of exposure group differences in the distribution of each covariate, and the association of covariates with the outcomes of interest was applied. The hazard ratio compare Empagliflozin versus Liraglutide (reference); Hazard Ratio (HR) = 1.01, 95% CI 2-sided [0.91 to 1.11] — Hazard ratio compares empagliflozin versus liraglutide (reference)

2. Primary Outcome: Incidence Rate of Expanded Major Adverse Cardiovascular Event (MACE) Composite Outcome - ITT Analysis
Description: Composite outcome includes: All-cause death, acute admission with non-fatal (within 30 days) stroke, with non-fatal (within 30 days) myocardial infarction (MI), admission with unstable angina, coronary revascularization, or acute admission with non-fatal heart failure (HF).
  The results from intention-to-treat (ITT) analysis are reported. For the ITT analyses, participants were defined as exposed from the start of treatment throughout follow-up, analogous to an ITT design in a interventional trial. Follow-up was not censored if glucose-lowering drugs other than the index drugs were prescribed in addition to empagliflozin or GLP-1RA after the index date.
Time Frame: From first initiation of empagliflozin or liraglutide until end of follow-up, up to 6 years.
Population: All patients included in the propensity score (PS) balanced cohort of either empagliflozin or liraglutide users.
Measure: Number; unit: Events per 1000 person-years
Arm/Group | Empagliflozin - PS Balanced Cohort | Liraglutide - PS Balanced Cohort
Number analyzed (Participants) | 14148 | 12626
Events per 1000 person-years | 39.9 | 37.3
Statistical Analysis 1: Comparison: Empagliflozin - PS Balanced Cohort vs Liraglutide - PS Balanced Cohort; Test type: Other — [test comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 1.07, 95% CI 2-sided [1.01 to 1.13] — Hazard ratio compares empagliflozin versus liraglutide (reference)

3. Secondary Outcome: Incidence Rate of Heart Failure (HF) Hospitalization or All-cause Death - OT Analysis
Description: The incidence rate of heart failure (HF) hospitalization or all-cause death based on on-treatment (OT) analysis is reported.
  For the OT analyses, treatment duration was based on the estimated number of days covered by each filled prescription, calculated as the number of drug packages times the numerical volume of a package. A grace period of 30 days were added.
  In the OT analysis, participants were censored from further follow-up at either treatment cessation, initiation of an alternative drug in the study drug class and initiation of a drug from the comparator study drug class.
Time Frame: From first initiation of empagliflozin or liraglutide until end of follow-up, up to 6 years.
Population: All patients included in the propensity score (PS) balanced cohort of either empagliflozin or liraglutide users.
Measure: Number; unit: Events per 1000 person-years
Arm/Group | Empagliflozin - PS Balanced Cohort | Liraglutide - PS Balanced Cohort
Number analyzed (Participants) | 14148 | 12626
Events per 1000 person-years | 21.1 | 22.2
Statistical Analysis 1: Comparison: Empagliflozin - PS Balanced Cohort vs Liraglutide - PS Balanced Cohort; Test type: Other — [test comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.95, 95% CI 2-sided [0.84 to 1.08] — Hazard ratio compares empagliflozin versus liraglutide (reference)

4. Secondary Outcome: Incidence Rate of Heart Failure (HF) Hospitalization or All-cause Death - ITT Analysis
Description: The incidence rate of heart failure (HF) hospitalization or all-cause death based on Intention-to-treat (ITT) analysis is reported. For the ITT analyses, participants are defined as exposed from the start of treatment throughout follow-up, analogous to an ITT design in a interventional trial. Follow-up was not censored if glucose-lowering drugs other than the index drugs were prescribed in addition to empagliflozin or GLP-1RA after the index date.
Time Frame: From first initiation of empagliflozin or liraglutide until end of follow-up, up to 6 years.
Population: All patients included in the propensity score (PS) balanced cohort of either empagliflozin or liraglutide users.
Measure: Number; unit: Events per 1000 person-years
Arm/Group | Empagliflozin - PS Balanced Cohort | Liraglutide - PS Balanced Cohort
Number analyzed (Participants) | 14148 | 12626
Events per 1000 person-years | 25.1 | 24.3
Statistical Analysis 1: Comparison: Empagliflozin - PS Balanced Cohort vs Liraglutide - PS Balanced Cohort; Test type: Other — [test comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 1.03, 95% CI 2-sided [0.96 to 1.11] — Hazard ratio compares empagliflozin versus liraglutide (reference)

5. Secondary Outcome: Incidence Rate of First Hospitalized Heart Failure (HHF) or Initiation of Community Prescription Drug Therapy With Loop Diuretics - OT Analysis
Description: The incidence rate of first hospitalized Heart Failure (HHF) or initiation of community prescription drug therapy with loop diuretics based on on-treatment (OT) analysis is reported.
  For the OT analyses, treatment duration was based on the estimated number of days covered by each filled prescription, calculated as the number of drug packages times the numerical volume of a package. A grace period of 30 days were added.
  In the OT analysis, participants were censored from further follow-up at either treatment cessation, initiation of an alternative drug in the study drug class and initiation of a drug from the comparator study drug class.
Time Frame: From first initiation of empagliflozin or liraglutide until end of follow-up, up to 6 years.
Population: All patients included in the propensity score (PS) balanced cohort of either empagliflozin or liraglutide users.
Measure: Number; unit: Events per 1000 person-years
Arm/Group | Empagliflozin - PS Balanced Cohort | Liraglutide - PS Balanced Cohort
Number analyzed (Participants) | 14148 | 12626
Events per 1000 person-years | 12.9 | 18.0
Statistical Analysis 1: Comparison: Empagliflozin - PS Balanced Cohort vs Liraglutide - PS Balanced Cohort; Test type: Other — [test comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.71, 95% CI 2-sided [0.61 to 0.83] — Hazard ratio compares empagliflozin versus liraglutide (reference)

6. Secondary Outcome: Incidence Rate of First Hospitalized Heart Failure (HHF) or Initiation of Community Prescription Drug Therapy With Loop Diuretics - ITT Analysis
Description: The incidence rate of first hospitalized Heart Failure (HHF) or initiation of community prescription drug therapy with loop diuretics based on intention-to-treat (ITT) analysis was reported. For the ITT analyses, participants are defined as exposed from the start of treatment throughout follow-up, analogous to an ITT design in a interventional trial. Follow-up was not censored if glucose-lowering drugs other than the index drugs were prescribed in addition to empagliflozin or GLP-1RA after the index date.
Time Frame: From first initiation of empagliflozin or liraglutide until end of follow-up, up to 6 years.
Population: All patients included in the propensity score (PS) balanced cohort of either empagliflozin or liraglutide users.
Measure: Number; unit: Events per 1000 person-years
Arm/Group | Empagliflozin - PS Balanced Cohort | Liraglutide - PS Balanced Cohort
Number analyzed (Participants) | 14148 | 12626
Events per 1000 person-years | 17.7 | 21.4
Statistical Analysis 1: Comparison: Empagliflozin - PS Balanced Cohort vs Liraglutide - PS Balanced Cohort; Test type: Other — [test comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.83, 95% CI 2-sided [0.76 to 0.91] — Hazard ratio compares empagliflozin versus liraglutide (reference)

7. Secondary Outcome: Incidence Rate of All-cause Hospitalization or Death - OT Analysis
Description: Incidence rate of all-cause hospitalization or death, based on on-treatment (OT) analysis is reported.
  For the OT analyses, treatment duration was based on the estimated number of days covered by each filled prescription, calculated as the number of drug packages times the numerical volume of a package. A grace period of 30 days were added. In the OT analysis, participants were censored from further follow-up at either treatment cessation, initiation of an alternative drug in the study drug class and initiation of a drug from the comparator study drug class.
Time Frame: From first initiation of empagliflozin or liraglutide until end of follow-up, up to 6 years.
Population: All patients included in the propensity score (PS) balanced cohort of either empagliflozin or liraglutide users.
Measure: Number; unit: Events per 1000 patient years
Arm/Group | Empagliflozin - PS Balanced Cohort | Liraglutide - PS Balanced Cohort
Number analyzed (Participants) | 14148 | 12626
Events per 1000 patient years | 193.5 | 212.1
Statistical Analysis 1: Comparison: Empagliflozin - PS Balanced Cohort vs Liraglutide - PS Balanced Cohort; Test type: Other — [test comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.92, 95% CI 2-sided [0.88 to 0.96] — Hazard ratio compares empagliflozin versus liraglutide (reference)

8. Secondary Outcome: Incidence Rate of All-cause Hospitalization or Death - ITT Analysis
Description: Incidence rate of all-cause hospitalization or death, based on intent-to-treat (ITT) analysis.
  For the ITT analyses, participants were defined as exposed from the start of treatment throughout follow-up, analogous to an ITT design in a interventional trial. Follow-up was not censored if glucose-lowering drugs other than the index drugs were prescribed in addition to empagliflozin or GLP-1RA after the index date.
Time Frame: From first initiation of empagliflozin or liraglutide until end of follow-up, up to 6 years.
Population: All patients included in the propensity score (PS) balanced cohort of either empagliflozin or liraglutide users.
Measure: Number; unit: Events per 1000 patient years
Arm/Group | Empagliflozin - PS Balanced Cohort | Liraglutide - PS Balanced Cohort
Number analyzed (Participants) | 14148 | 12626
Events per 1000 patient years | 175.2 | 187.0
Statistical Analysis 1: Comparison: Empagliflozin - PS Balanced Cohort vs Liraglutide - PS Balanced Cohort; Test type: Other — [test comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.94, 95% CI 2-sided [0.91 to 0.96] — Hazard ratio compares empagliflozin versus liraglutide (reference)

9. Secondary Outcome: Incidence Rate of All Cause Hospitalization - OT Analysis
Description: Incidence rate of all cause hospitalization, based on on-treatment (OT) analysis is reported.
  For the OT analyses, treatment duration was based on the estimated number of days covered by each filled prescription, calculated as the number of drug packages times the numerical volume of a package. A grace period of 30 days were added. In the OT analysis, participants were censored from further follow-up at either treatment cessation, initiation of an alternative drug in the study drug class and initiation of a drug from the comparator study drug class.
Time Frame: From first initiation of empagliflozin or liraglutide until end of follow-up, up to 6 years.
Population: All patients included in the propensity score (PS) balanced cohort of either empagliflozin or liraglutide users.
Measure: Number; unit: Events per 1000 patient years
Arm/Group | Empagliflozin - PS Balanced Cohort | Liraglutide - PS Balanced Cohort
Number analyzed (Participants) | 14148 | 12626
Events per 1000 patient years | 190.2 | 208.0
Statistical Analysis 1: Comparison: Empagliflozin - PS Balanced Cohort vs Liraglutide - PS Balanced Cohort; Test type: Other — [test comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.92, 95% CI 2-sided [0.88 to 0.96] — Hazard ratio compares empagliflozin versus liraglutide (reference)

10. Secondary Outcome: Incidence Rate of All Cause Hospitalization - ITT Analysis
Description: Incidence rate of all cause hospitalization, based on intent-to-treat (ITT) analysis.
  For the ITT analyses, participants were defined as exposed from the start of treatment throughout follow-up, analogous to an ITT design in a interventional trial. Follow-up was not censored if glucose-lowering drugs other than the index drugs were prescribed in addition to empagliflozin or GLP-1RA after the index date.
Time Frame: From first initiation of empagliflozin or liraglutide until end of follow-up, up to 6 years.
Population: All patients included in the propensity score (PS) balanced cohort of either empagliflozin or liraglutide users.
Measure: Number; unit: Events per 1000 patient years
Arm/Group | Empagliflozin - PS Balanced Cohort | Liraglutide - PS Balanced Cohort
Number analyzed (Participants) | 14148 | 12626
Events per 1000 patient years | 171.6 | 183.7
Statistical Analysis 1: Comparison: Empagliflozin - PS Balanced Cohort vs Liraglutide - PS Balanced Cohort; Test type: Other — [test comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.93, 95% CI 2-sided [0.91 to 0.96] — Hazard ratio compares empagliflozin versus liraglutide (reference)

11. Secondary Outcome: Incidence Rate of All-cause Death - OT Analysis
Description: Incidence rate of all-cause death, based on on-treatment (OT) analysis is reported.
  For the OT analyses, treatment duration was based on the estimated number of days covered by each filled prescription, calculated as the number of drug packages times the numerical volume of a package. A grace period of 30 days were added.
  In the OT analysis, participants were censored from further follow-up at either treatment cessation, initiation of an alternative drug in the study drug class and initiation of a drug from the comparator study drug class.
Time Frame: From first initiation of empagliflozin or liraglutide until end of follow-up, up to 6 years.
Population: All patients included in the propensity score (PS) balanced cohort of either empagliflozin or liraglutide users.
Measure: Number; unit: Events per 1000 patient-years
Arm/Group | Empagliflozin - PS Balanced Cohort | Liraglutide - PS Balanced Cohort
Number analyzed (Participants) | 14148 | 12626
Events per 1000 patient-years | 12.9 | 13.2
Statistical Analysis 1: Comparison: Empagliflozin - PS Balanced Cohort vs Liraglutide - PS Balanced Cohort; Test type: Other — [test comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.99, 95% CI 2-sided [0.83 to 1.18] — Hazard ratio compares empagliflozin versus liraglutide (reference)

12. Secondary Outcome: Incidence Rate of All-cause Death - ITT Analysis
Description: Incidence rate of all-cause death, based on intent-to-treat (ITT) analysis. For the ITT analyses, participants were defined as exposed from the start of treatment throughout follow-up, analogous to an ITT design in a interventional trial. Follow-up was not censored if glucose-lowering drugs other than the index drugs were prescribed in addition to empagliflozin or GLP-1RA after the index date.
Time Frame: From first initiation of empagliflozin or liraglutide until end of follow-up, up to 6 years.
Population: All patients included in the propensity score (PS) balanced cohort of either empagliflozin or liraglutide users.
Measure: Number; unit: Events per 1000 patient-years
Arm/Group | Empagliflozin - PS Balanced Cohort | Liraglutide - PS Balanced Cohort
Number analyzed (Participants) | 14148 | 12626
Events per 1000 patient-years | 18.0 | 17.1
Statistical Analysis 1: Comparison: Empagliflozin - PS Balanced Cohort vs Liraglutide - PS Balanced Cohort; Test type: Other — [test comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 1.06, 95% CI 2-sided [0.97 to 1.16] — Hazard ratio compares empagliflozin versus liraglutide (reference)

13. Secondary Outcome: Incidence Rate of Hospitalization for Heart Failure (HF) - OT Analysis
Description: Incidence rate of hospitalization for heart failure (HF), based on on-treatment (OT) analysis is reported.
  For the OT analyses, treatment duration was based on the estimated number of days covered by each filled prescription, calculated as the number of drug packages times the numerical volume of a package. A grace period of 30 days were added.
  In the OT analysis, participants were censored from further follow-up at either treatment cessation, initiation of an alternative drug in the study drug class and initiation of a drug from the comparator study drug class.
Time Frame: From first initiation of empagliflozin or liraglutide until end of follow-up, up to 6 years.
Population: All patients included in the propensity score (PS) balanced cohort of either empagliflozin or liraglutide users.
Measure: Number; unit: Events per 1000 patient years
Arm/Group | Empagliflozin - PS Balanced Cohort | Liraglutide - PS Balanced Cohort
Number analyzed (Participants) | 14148 | 12626
Events per 1000 patient years | 9.3 | 10.6
Statistical Analysis 1: Comparison: Empagliflozin - PS Balanced Cohort vs Liraglutide - PS Balanced Cohort; Test type: Other — [test comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.87, 95% CI 2-sided [0.72 to 1.06] — Hazard ratio compares empagliflozin versus liraglutide (reference)

14. Secondary Outcome: Incidence Rate of Hospitalization for Heart Failure (HF) - ITT Analysis
Description: Incidence rate of hospitalization for heart failure (HF), based on intent-to-treat (ITT) analysis.
  For the ITT analyses, participants were defined as exposed from the start of treatment throughout follow-up, analogous to an ITT design in a interventional trial. Follow-up was not censored if glucose-lowering drugs other than the index drugs were prescribed in addition to empagliflozin or GLP-1RA after the index date.
Time Frame: From first initiation of empagliflozin or liraglutide until end of follow-up, up to 6 years.
Population: All patients included in the propensity score (PS) balanced cohort of either empagliflozin or liraglutide users.
Measure: Number; unit: Events per 1000 patient years
Arm/Group | Empagliflozin - PS Balanced Cohort | Liraglutide - PS Balanced Cohort
Number analyzed (Participants) | 14148 | 12626
Events per 1000 patient years | 9.3 | 9.4
Statistical Analysis 1: Comparison: Empagliflozin - PS Balanced Cohort vs Liraglutide - PS Balanced Cohort; Test type: Other — [test comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.98, 95% CI 2-sided [0.88 to 1.10] — Hazard ratio compares empagliflozin versus liraglutide (reference)

ADVERSE EVENTS:
Time Frame: From first initiation of empagliflozin or liraglutide until end of follow-up, up to 6 years.
Description: This is a non-interventional study using electronic health care records, with data retrieved from Danish National Patient Registry, Danish National Prescription Registry and Danish Register of Causes of Death. No adverse events were collected on an individual case level. "0" in the Serious Adverse Events, and Other Adverse Events parts refer to not applicable.
  All-cause death for ITT analysis is reported.
Arm/Group | Empagliflozin - PS Balanced Cohort | Liraglutide - PS Balanced Cohort
All-Cause Mortality (participants affected / at risk) | 881/14148 | 765/12626
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Due to a huge shift after 2018 in drug type use within the GLP-1RA group the final analysis (between 2015 - 2020) was not completed. Instead, an exploratory analysis was performed, using the initial analysis of comparing from empagliflozin versus liraglutide from 2015 to 2018 but following these same patients up to 2020.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results.

Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days.

BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-11-08): https://cdn.clinicaltrials.gov/large-docs/32/NCT03993132/Prot_SAP_000.pdf